CLINICAL TRIAL: NCT03745079
Title: Correlation Between Core Temperature and Skin Temperature Measured by 3M SpotOn
Acronym: Temperature
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ajou University School of Medicine (Other)
Responsible Party: Principal Investigator, In-kyong Yi, Clinical assistant professor, Ajou University School of Medicine
Other Study IDs: MED-OBS-18-350
Record Dates: First submitted 2018-11-12; First posted 2018-11-19 (Actual); Last update posted 2023-03-06 (Actual); Status verified 2023-03

CONDITIONS: Temperature; General Anesthesia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group 1: Participants' temperature measured at 3 places at the same time
  * Esophagus
  * Skin near to temporal artery
  * Skin near to carotid artery
  Interventions: Other: Esophagus temperature monitoring; Other: Spoton Temporal; Other: Spoton Carotid

INTERVENTIONS:
Other: Esophagus temperature monitoring — Measuring core temperature by esophageal stethoscope
  Other Names: Core temperature
Other: Spoton Temporal — Mesuring temperature on skin near to temporal artery using Spoton
  Other Names: Mesuring temperature on skin near to temporal artery
Other: Spoton Carotid — Mesuring temperature on skin near to carotidl artery using Spoton
  Other Names: Mesuring temperature on skin near to carotid artery

SUMMARY:
Core temperature should be monitored under general anesthesia. Recently developed 3M Spoton skin temeprature which is applied on temporal artery is correlated with core temperature measure by esophageal prove in several studies. Conventional skin temperature over carotid artery is also correlated with core temperature in several studies. The purpose of this study is comparing 3 methods of temperature monitoring. First, conventional core temperature measure by esophageal stethoscope. Second, 3M Spoton applying on temporal artery. Third, 3M Spoton applying on carotid artery

DETAILED DESCRIPTION:
Core temperature should be monitored under general anesthesia. Because patients are prone to hypothermia during surgery. Conventional core temperature is monitored at esophagus, rectum, nasopharynx. But some of them are invasive and impossible in sometimes. Recently developed 3M Spoton skin temeprature which is applied on temporal artery is correlated with core temperature measured by esophageal prove in several studies. Its mechanism is making zero heat flux on skin applied. But it also cannot apply in head or facial surgery. Other studies showed conventional skin temperature over carotid artery is also correlated with core temperature. The investigators hypothesized using Spoton on carotid artery could be alternative method measuring core temperature. The purpose of this study is comparing 3 methods of temperature monitoring. First, conventional core temperature measure by esophageal stethoscope. Second, 3M Spoton applying on temporal artery. Third, 3M Spoton applying on carotid artery

ELIGIBILITY:
Inclusion Criteria:

* Age 19~60 years old
* Who need surgery more than 2 hours under general anesthesia
* American Society of Anesthesiologists physical status 1 or 2

Exclusion Criteria:

* Body mass index < 35
* Head and neck surgery
* Patients with fever > 38'C
* History of malignant hyperthermia

Ages: 19 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients who scheduled surgery more than 2 hours under general anesthesia. Who need esophageal temperature monitoring for routine monitoring.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2019-09-20 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Esophageal core temperature measured by stethoscope ℃ | 3 hours (during general anesthesia)
  Temperature measured by esophageal stethoscope, ℃
Carotid skin temperature by SpotOn, ℃ | 3 hours (during general anesthesia)
  Temperature measured by SpotOn near to carotid artery, ℃
Temporal skin temperature by SpotOn, ℃ | 3 hours (during general anesthesia)
  Temperature measured by SpotOn near to temporal artery, ℃

SECONDARY OUTCOMES:
Room temperature, ℃ | 3 hours (during general anesthesia)
  Operating room temperature, ℃

CONTACTS AND LOCATIONS:
Overall Officials: In Kyong Yi, MD, Principal Investigator — Ajou University School of Medicine
Locations (1):
- Ajou university school of medicine, Suwon, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: Undecided